CLINICAL TRIAL: NCT02720952
Title: A Phase 3 Open-label Study of Infacort® in Neonates, Infants and Children Less Than 6 Years of Age With Adrenal Insufficiency
Brief Title: Treatment of Adrenal Insufficiency in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Treatment of Adrenal Insufficiency in Neonates consortium (TAIN) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Infacort-003
Record Dates: First submitted 2016-03-16; First posted 2016-03-28 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infacort (Experimental): Infacort® is a dry granule formulation of hydrocortisone stored in capsules that will be available in different strengths (0.5, 1.0, 2.0 and 5.0mg).
  The clinically-appropriate dose, based on standard individualised treatment, will be administered, given as a single dose orally. This will usually be equivalent to the previous day's dose.
  Interventions: Drug: Infacort®

INTERVENTIONS:
Drug: Infacort® — dry granule formulation of hydrocortisone

SUMMARY:
The study will be conducted in a total of 24 subjects before their 6th birthday, requiring replacement therapy for adrenal insufficiency due to either CAH, primary adrenal failure or hypopituitarism.

The study will consist of three consecutive cohorts. Cohort 1 will include 12 subjects aged between 2 and < 6 years. If no safety concerns emerge, then 6 subjects aged 28 days to <2 years will be enrolled (Cohort 2). A review of accumulated data will be undertaken and only if again no safety concerns emerge, then 6 neonates aged from birth to <28 days will be enrolled (Cohort 3).

The decision to continue after each cohort will be based on the recommendation of an Independent Data Monitoring Committee (IDMC).

DETAILED DESCRIPTION:
This is a Phase 3, open label, single centre study of Infacort® in neonates, infants and children less than 6 years of age with adrenal insufficiency. The study will be conducted in a total of 24 subjects, before their 6th birthday, requiring replacement therapy for adrenal insufficiency due to either CAH, primary adrenal failure or hypopituitarism. Due to the rare occurrence of adrenal insufficiency it is expected that for the third cohort of this study (neonates) only subjects with CAH will be recruited.

The study will consist of three consecutive parts. Cohort 1 will include 12 subjects aged between 2 and < 6 years. If no safety concerns emerge, then 6 subjects aged 28 days to <2 years will be enrolled (Cohort 2). A review of accumulated data will be undertaken and only if again no safety concerns emerge, then 6 neonates aged from birth to <28 days will be enrolled (Cohort 3).

The decision to continue after each cohort will be based on the recommendation of an Independent Data Monitoring Committee (IDMC).

The study will consist of a screening visit (Visit 1 performed as a minimum the day before the intake of study drug), one treatment visit (Visit 2, Day 1), a follow-up visit (Visit 3) one to three days after intake of study drug (Day 2, Day 3 or Day 4) and a follow-up telephone call (Visit 4) 7 - 10 days after intake of study drug. Study completion evaluation will be performed at Visit 3. Parents/ carers will have at least 1 night to consider participation of their child before completing written informed consent. Children aged 3 - 6 years will be informed about their involvement in the study in the presence of their parents/carers.

All subjects will receive their standard treatment including fludrocortisone other than the dose of hydrocortisone that is to be substituted by Infacort®.

Subjects who meet the eligibility criteria at screening (Visit 1) will attend for Visit 2 at a suitable time before the next planned dose of hydrocortisone is due. Subjects may have insertion of an intravenous cannula (with suitable local anaesthesia) allowing blood samples to be taken as well as their routine clinical samples (where required) prior to their next dose of hydrocortisone given as Infacort®. If a cannula is not used, direct venous sampling may be carried out instead. After all planned study procedures have been completed the subjects will go home and will return one to three days later for the follow-up assessments (Visit 3). A follow-up telephone call (Visit 4) 7 - 10 days after intake of study drug will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female children less than 6 years of age.
2. A diagnosis of adrenal insufficiency as confirmed by an inappropriately low cortisol usually with other supporting tests.
3. Receiving appropriate adrenocortical replacement therapy (hydrocortisone with/without fludrocortisone).
4. Adequately hydrated and nourished.
5. Ability of parents/carers to understand and give written Informed Consent

Exclusion Criteria:

1. Clinically evident acute adrenal insufficiency (adrenal crisis).
2. Inability of the child to take oral therapy.
3. Concomitant therapy (other than that required to treat adrenal insufficiency, Vitamin D, Fluoride, Thyroxine and growth hormone).
4. Subjects with clinical signs of acute infection or fever on Day 1.
5. Any surgical or medical condition which in the opinion of the investigator may place the subject at higher risk from his/her participation in the study.
6. Parents/carers of subjects unwilling to consent to saving and propagation of pseudonymised medical data for study reasons.
7. Subjects who are dependent on the investigator or the sponsor.

Ages: 1 Week to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Wiegand, MD, Principal Investigator — Charité-Universitätsmedizin Berlin, CVK
Locations (1):
- Charité-Universitätsmedizin Berlin, CVK, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Infacort: Infacort® is a dry granule formulation of hydrocortisone stored in capsules that will be available in different strengths (0.5, 1.0, 2.0 and 5.0mg).
  The clinically-appropriate dose, based on standard individualised treatment, will be administered, given as a single dose orally. This will usually be equivalent to the previous day's dose.
  Infacort®: dry granule formulation of hydrocortisone
Period: Overall Study
Arm/Group | Infacort
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infacort
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: days] | 718.1 [16 to 1708]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 24

OUTCOME MEASURES:

1. Primary Outcome: Serum Cortisol Concentration up to 240 Minutes
Description: The primary endpoint will be the maximum levels of serum cortisol concentration up to 240 minutes after intake of study drug as determined by the central laboratory.
Time Frame: 240 minutes
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Infacort
Number analyzed (Participants) | 24
nmol/L | 575.8 (47.9)

2. Secondary Outcome: Serum Cortisol Concentration up to 6 Hours
Description: Serum cortisol concentration 240 minutes after intake of study drug as determined by the central laboratory
Time Frame: 240 minutes
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Infacort
Number analyzed (Participants) | 24
nmol/L | 60.1 (131.7)

3. Secondary Outcome: Subject Assessment of Taste of the Product
Description: Palatability of the investigational product as determined by parent/carer responses to the following questions:
  Question 1: My child found swallowing easy. Question 2: My child showed a positive reaction after Infacort was given. Question 3: I would be happy to give my child Infacort in the future. Question 4: Overall, I would prefer Infacort for my child over the usual hydrocortisone medication.
Time Frame: 1 minute
Population: Out of the total population, one parent/carer did not complete the palatability questionnaire and one parent/carer did not complete questions 3 and 4, and thus were excluded from the analysis of the relevant questions.
Measure: Count of Participants; unit: Participants
Groups:
- Question 1: Percentage of parents/carers that agreed, or strongly agreed with the statement: My child found swallowing easy.
- Question 2: Percentage of parents/carers that agreed, or strongly agreed with the statement: My child showed a positive reaction after Infacort was given.
- Question 3: Percentage of parents/carers that agreed, or strongly agreed with the statement: I would be happy to give my child Infacort in the future.
- Question 4: Percentage of parents/carers that agreed, or strongly agreed with the statement: Overall, I would prefer Infacort for my child over the usual hydrocortisone medication.
Arm/Group | Question 1 | Question 2 | Question 3 | Question 4
Number analyzed (Participants) | 23 | 23 | 22 | 22
Participants | 19 | 15 | 21 | 21

4. Secondary Outcome: Incidence of Serious Adverse Events (SAEs) and Adverse Events (AE)
Description: Incidence of serious adverse events (SAEs) and adverse events (AE).
Time Frame: 7-10 days
Measure: Number; unit: Adverse Events
Arm/Group | Infacort
Number analyzed (Participants) | 24
Adverse Events
  Treatment-Emergent | 12
  Serious TEAEs | 0
  Severe TEAEs | 0
  Moderate TEAEs | 2
  Mild TEAEs | 10

ADVERSE EVENTS:
Description: Adverse Events will be recorded from the time of first intake of Infacort® until Visit 4. Serious Adverse Events (SAEs) will be recorded from the time of first intake of Infacort® until 7 days following administration of Infacort®. Any SAEs experienced after this 7-day period will be reported to the sponsor if the investigator suspects a causal relationship to the study drug.
Arm/Group | Infacort
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 8/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infacort (N=24)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Infantile spitting up (Gastrointestinal disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No